CLINICAL TRIAL: NCT03071081
Title: A Phase 1 Study to Evaluate the Safety, Tolerability and Pharmacokinetics of TOP1288 Oral Single Ascending and Multiple Doses in Healthy Volunteers
Brief Title: Study for Safety and Tolerability of TOP1288 Administered Orally in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Topivert Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TOP1288-TV-03
Record Dates: First submitted 2017-02-20; First posted 2017-03-06 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: 3 dose groups (2 arms per dose group)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- TOP1288 200mg BID (Experimental): 1 day dosing
  Interventions: Drug: TOP1288
- Placebo to TOP1288 200mg BID (Placebo Comparator): 1 day dosing
  Interventions: Drug: Placebo to TOP1288
- TOP1288 1g BID (Experimental): 1 day dosing
  Interventions: Drug: TOP1288
- Placebo to TOP1288 1g BID (Placebo Comparator): 1 day dosing
  Interventions: Drug: Placebo to TOP1288
- TOP1288 Xg (where X is <=1g) BID (Experimental): 7 days dosing
  Interventions: Drug: TOP1288
- Placebo to TOP1288 Xg (Placebo Comparator): 7 days dosing
  Interventions: Drug: Placebo to TOP1288

INTERVENTIONS:
Drug: TOP1288 — Oral TOP1288
  Arms: TOP1288 1g BID; TOP1288 200mg BID; TOP1288 Xg (where X is <=1g) BID
Drug: Placebo to TOP1288 — Oral placebo to TOP1288
  Arms: Placebo to TOP1288 1g BID; Placebo to TOP1288 200mg BID; Placebo to TOP1288 Xg

SUMMARY:
This study evaluates the safety and tolerability of TOP1288 oral single ascending and multiple doses in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a healthy male, aged between 18 and 55 years of age (inclusive) at Screening.
2. Subject has a body mass index (BMI) of between 18.0 and 29.9 kg/m2 (inclusive), with a body weight of at least 50 kg at Screening.
3. Subject is in good physical and mental health in the opinion of the Investigator.
4. Subject has clinical laboratory test results within the reference ranges of the testing laboratory unless results outside the reference ranges are deemed not clinically significant by the Investigator at Screening and Day -1.
5. Subject has a supine blood pressure and pulse rate within the normal range after 5 minutes' rest (systolic blood pressure: 90 to 140 mmHg, diastolic blood pressure: 40 to 90 mmHg, pulse rate: 40 to 90 beats per minute) at Screening and Day -1.
6. Subjects must be willing to comply with the contraception restrictions of the protocol for this study.
7. Subject has regular bowel opening of usually 1 motion per day of normal consistency.

Exclusion Criteria:

1. Subject has participated in another study of an investigational medication (or a medical device) within the last 3 months or 5 half-lives of the investigational medication, whichever is longer, prior to the first day or dosing.
2. Subject has made a blood donation (> 400 mL) or had a comparable blood loss (> 350 mL) within the last 3 months prior to first administration of study drug.
3. Subject tests positive for human immunodeficiency virus (HIV)-1/2 antibodies, hepatitis B surface antigen, or hepatitis C antibodies at Screening.
4. Subject has a history of alcohol and/or drug abuse.
5. Subject has an alcohol consumption of more than 21 units of alcohol per week.
6. Subject tests positive for alcohol and/or drugs (urine tests) at Screening or admission.
7. Subject has received any prescription or non-prescription medications, including over-the-counter medications, nutraceuticals (e.g., St. John's Wort, ginseng, kava kava, Ginkgo biloba and melatonin), foods or beverages containing grapefruit and vitamin supplements within 14 days prior to admission (Day -1) or nutraceuticals containing caffeine- or xanthine-related substances within 72 hours prior to admission (Day -1). Foods or beverages containing Seville-type (sour) oranges, or poppy seeds are also excluded within this time period.
8. The subject has a history of daily consumption of 5 or more cups of coffee or tea.
9. Subject has a known hypersensitivity to any components of the study drug.
10. Subject has any history of any clinically significant acute or chronic condition affecting the colon and/or rectum and/or anus, including haemorrhoids and irritable bowel syndrome, sufficient to cause symptoms and/or that in the judgement of the PI and the Sponsor's study Physician/Medical Monitor would interfere with the subject's participation in the study.
11. Any findings on pre-dose endoscopy that in the PI's judgement would interfere with subject participation in the study.
12. Subject has acute or chronic condition affecting GI motility such as constipation or diarrhoea that would, in the judgement of the PI and the Sponsor's study Physician/Medical Monitor, interfere with the subject's participation in the study
13. Subject has cardiovascular or cerebrovascular disease, including hypertension, angina, ischaemic heart disease, transient ischaemic attacks, stroke and peripheral arterial disease sufficient to cause symptoms and/or require therapy to maintain stable status.
14. Subject has an active infection (e.g., sepsis, pneumonia, abscess) or has had a serious infection (resulting in hospitalisation or requiring parenteral antibiotic treatment) within 6 weeks prior to study drug administration.
15. Subject has a history of positive tuberculosis test or evidence of possible tuberculosis or latent tuberculosis infection at Screening (interferon gamma release assay testing) that cannot be attributed to a prior Bacillus Calmette-Guérin inoculation.
16. Subject has received live attenuated vaccination within 6 weeks prior to Screening or intends to have such a vaccination during the course of the study.
17. Subject has any of the following haematology values at Screening or Day -1:

    * Haemoglobin, < 13 g/dL.
    * Absolute neutrophil count < 1.5 x 109/L (< 1500/μL).
18. Subject has a 12-lead electrocardiogram (ECG) with results considered to be potentially clinically significant, e.g., QTcF > 450 ms, bundle branch block, evidence of myocardial ischaemia, at Screening or Day -1.
19. Subject has an abnormality in the ECG that, in the opinion of the Investigator, increases the risks associated with participating in the study.
20. Subject has renal or liver impairment at Screening or Day -1, defined as:

    * Serum creatinine level ≥ 135 μmol/L, or
    * Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≥2 x upper limit of normal, or
    * Alkaline phosphate and/or bilirubin > 1.5 x upper limit of normal (an isolated bilirubin 1.5 x upper limit of normal is acceptable if bilirubin is fractionated and direct bilirubin is < 35%).
21. Subject has active neoplastic disease or history of any neoplastic disease within 5 years of Screening (except for basal or squamous cell carcinoma of the skin or carcinoma in situ that has been definitively treated with standard of care).
22. Subject has any other acute or chronic illness which, in the opinion of the Investigator or Sponsor's study Physician/Medical Monitor, could pose a threat or harm to the subject's participation in the study.
23. The subject has used nicotine-containing products (including, but not limited to, cigarettes, pipes, cigars, chewing tobacco, nicotine patch, or nicotine gum) within 2 weeks prior to admission to the study centre (Day -1).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-06-02 (Actual)

PRIMARY OUTCOMES:
Safety (AEs) | To 7 days after last dose
  As measured by adverse events
Safety (ECGs) | To 7 days after last dose
  As measured by ECGs
Safety (vital signs) | To 7 days after last dose
  As measured by vital signs
Safety (clinical lab tests) | To 7 days after last dose
  As measured by clinical laboratory tests

SECONDARY OUTCOMES:
Pharmacokinetic profile Cmax | 0-48 hours
  Observed maximum plasma concentration, taken directly from the individual concentration-time curve (Cmax)
Pharmacokinetic profile AUC | 0-48 hours
  Area under the plasma concentration-curve (AUC)
Pharmacokinetic profile AUC0-12h | 0-12 hours
  AUC from time zero to 12 h (AUC0-12h)
Pharmacokinetic profile AUC0-24h | 0-24 hours
  AUC from time zero to 24 h (AUC0-24h)
Pharmacokinetic profile AUC0-t | 0-48 hours
  AUC from time zero to the last measurable concentration (AUC0-t)
Pharmacokinetic profile Racc | 0-48 hours
  Accumulation ratio of the AUC (Racc) (multiple dose part only)
Pharmacokinetic profile tmax | 0-48 hours
  Time to reach maximum concentration, taken directly from the individual concentration-time curve (tmax)
Pharmacokinetic profile t½ | 0-48 hours
  Terminal half-life (t½)
Pharmacokinetic profile λz | 0-48 hours
  Terminal elimination rate constant (λz)
Pharmacokinetic profile CL/F | 0-48 hours
  Apparent total clearance from plasma after oral administration (CL/F)
Pharmacokinetic profile Vz/F | 0-48 hours
  Volume of distribution of the absorbed fraction (Vz/F)

CONTACTS AND LOCATIONS:
Overall Officials: Muna Albayaty, MBChB, FFPM, Principal Investigator — Copenhagen Trial Unit, Center for Clinical Intervention Research
Locations (1):
- PAREXEL Early Phase Clinical Unit, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No